CLINICAL TRIAL: NCT05404711
Title: Feasibility and Acceptability of Home Use Continuous Glucose Monitors for Type 2 Diabetes Risk Evaluation in Youth
Brief Title: Continuous Glucose Monitors (CGM) for Type 2 Diabetes (T2D) Risk Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Ellen Vajravelu, MD (Other)
Responsible Party: Sponsor-Investigator, Mary Ellen Vajravelu, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY22030082
Record Dates: First submitted 2022-05-25; First posted 2022-06-03 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity; PreDiabetes; Insulin Resistance
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Subjects will wear a continuous glucose monitor (CGM) to determine the feasibility and acceptability of the device to evaluate risk of youth developing Type 2 Diabetes (T2D).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM use for T2D risk evaluation (Other): All participants will complete a standard 2-hour oral glucose tolerance test (OGTT), wear a CGM for 10 days, complete at-home glucose challenge, and provide qualitative feedback about their experiences with both OGTT and CGM use for risk evaluation.
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Participants will wear blinded Dexcom G6 Pro continuously for 10 days in their home environment. Two challenges will be completed at home: 1) glucose, using 1.75 g/kg (max 75g) glucose beverage provided by study team, and 2) mixed food, containing 50g carb as well as protein and fat content of participant's choice.

SUMMARY:
The purpose of this research study is to determine whether continuous glucose monitors (CGM) are a safe, effective, and acceptable way to evaluate type 2 diabetes risk in youth as compared to the standard 2-hour oral glucose tolerance test (OGTT).

This study will involve wearing a CGM, wearing a physical activity tracker, responding to surveys, and completing at-home glucose and mixed food challenge while wearing the CGM. Subjects will also be asked to complete an interview by phone or videoconference after wearing the CGM.

DETAILED DESCRIPTION:
Youth-onset type 2 diabetes (T2D), an increasingly common and aggressive disease that disproportionately impacts racial and ethnic minorities, presents several diagnostic challenges. The rapid loss of glycemic control soon after T2D diagnosis makes early identification an important goal in pediatrics, and risk-based screening has been recommended for children for over two decades. However, the screening tests currently used in practice, including hemoglobin A1c (HbA1c), fasting glucose, and 2-hour oral glucose tolerance test (OGTT), have significant drawbacks. Real-time continuous glucose monitors (CGM) are promising new tools for risk stratification in individuals with dysglycemia. These patient-worn medical devices measure interstitial glucose every 5 minutes and offer glimpses into an individual's everyday life, which may include consumption of carbohydrates in amounts larger than that assessed in an OGTT, enhancing test sensitivity. Whether use of CGMs to evaluate type 2 diabetes risk in free-living youth is feasible and acceptable to patients and families is unknown. Assessment of CGM with standardized, but practical, home-based glucose and mixed-meal challenges is needed to determine facilitators and barriers to use of this technology-driven approach in clinical practice. Without advancement in the approach to screening for youth-onset T2D, there is ongoing risk of failure to understand which individuals are at highest risk for complications and could benefit the most from intervention early in the disease process.

In this single-arm prospective study, participants will attend one in-person study visit to complete 2-hour oral glucose tolerance test after overnight fast. Participants will wear a continuous glucose monitor and a wrist-worn actigraphy device for physical activity and sleep measurement for 10 days beginning on the day of the study visit, then return the monitors by mail. During the 10 day wear period, participants will respond to text message-based surveys to document food intake, physical activity, and sleep times and will complete two at-home challenges: 1) glucose challenge using study-provided glucose beverage that is identical to that they consume during clinical oral glucose tolerance test; and 2) food challenge with mixed carbohydrate/fat/protein-containing food of their choice. Glucose trends during these at-home challenges will be compared with oral glucose tolerance test obtained during the study visit. Individual interviews will be conducted upon completion of CGM wear to assess acceptability of the use of at-home glucose challenge and CGM wear as a strategy to evaluate diabetes risk in youth.

ELIGIBILITY:
Inclusion Criteria:

* Any gender, age 8-18 years
* Tanner 2 or higher pubertal development
* Overweight or obese (BMI ≥85th percentile for age/sex, or ≥ 25 kg/m2 for participants =18 years)
* A) No previously documented abnormal HbA1c or glucose but at higher risk for T2D based on race/ethnicity (Black, Hispanic, Asian, Native American, Pacific Islander), diagnosis with dyslipidemia, hypertension, polycystic ovary syndrome, presence of acanthosis nigricans, or first degree relative with T2D; or B) previously documented (within 6 months) HbA1c 5.7-7.0%, fasting glucose ≥100 mg/dL, or 2-hour plasma glucose on OGTT of ≥140 mg/dL
* Consent (adult subjects), parental/guardian permission (if applicable), assent (if applicable)
* Willingness to wear ActiGraph watch and CGM continuously for 10 day study duration

Exclusion Criteria:

* Current or recent (within 1 month) use of diabetes-related medication
* Current use of hydroxyurea (due to interference with CGM)
* Known type 1, cystic fibrosis-related, or medication-induced diabetes
* Potential subject unable to speak or read in English
* Severe cognitive impairment
* Current or previous pregnancy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen Vajravelu, MD, MSHP, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Completed Study Visit
Arm/Group | CGM Use for T2D Risk Evaluation
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Completed 75-gram, 2-hour CGM-OGTT
Arm/Group | CGM Use for T2D Risk Evaluation
Started | 39
Completed | 35
Not Completed | 4
Not completed — Incomplete due to illness | 1
Not completed — CGM fell off early | 3
Period: Valid 75-gram, 2-hour CGM-OGTT
Arm/Group | CGM Use for T2D Risk Evaluation
Started | 35
Completed | 30
Not Completed | 5
Not completed — No date/time recorded | 4
Not completed — Vomited after drinking glucose beverage at home | 1
Period: Completed, Valid Lab-OGTT and CGM-OGTT
Arm/Group | CGM Use for T2D Risk Evaluation
Started | 30
Completed | 29
Not Completed | 1
Not completed — Incomplete glucose beverage for lab-OGTT | 1

BASELINE CHARACTERISTICS:
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.6 [12.9 to 16.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: non-Hispanic White | 18
  Race/Ethnicity: non-Hispanic Black | 13
  Race/Ethnicity: multi-racial | 5
  Race/Ethnicity: Hispanic/Latinx | 3
Region of Enrollment [Number; unit: participants]
  United States | 39
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 35.9 [31.7 to 41.0]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of CGM Use to Determine Type 2 Diabetes Risk
Description: Completeness of CGM data (≥ 80% of days with data)
Time Frame: 10 days
Population: Of the 39 participants who completed the study visit, 38 returned their CGM for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 38
Participants
  CGM Wear ≥ 8 Days | 33
  CGM Wear < 8 Days | 5

2. Secondary Outcome: Acceptability of CGM Use for At-home T2D Risk Evaluation in Youth
Description: Interview-based assessment. Participants rated their experience with CGM-OGTT using a Likert-like scale from 1-5 (1= terrible, 2=bad, 3=neutral, 4=good, 5=excellent). Acceptability was defined as a pre-specified threshold of ≥80% of participants providing a neutral or higher rating.
Time Frame: 30 minutes
Population: Of the 39 participants enrolled in the study, only 36 completed the exit interview.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 36
Participants
  Rated as excellent/good | 33
  Rated as neutral | 3

3. Secondary Outcome: Sensitivity of At-home CGM-measured Glucose Challenge
Description: Sensitivity of CGM-glucose 2 hours after at-home glucose beverage ingestion to predict OGTT-2h≥140 mg/dL
Time Frame: 2 Hour Point of Home-OGTT
Measure: Number; unit: percentage of true positives
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 29
percentage of true positives | 80
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 0.56, 95% CI 2-sided [0.18 to 0.94] — Area under the receiver operating characteristic curve (AUC) was 0.56 (95% CI 0.18-0.94) for 2-hour postprandial glucose

4. Secondary Outcome: Specificity of At-home CGM-measured Glucose Challenge
Description: Specificity of CGM-glucose 2 hours after at-home glucose beverage ingestion to predict OGTT-2h≥140 mg/dL
Time Frame: 2 Hour Point of Home-OGTT
Measure: Number; unit: percentage of true negatives
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 29
percentage of true negatives | 25
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 0.56, 95% CI 2-sided [0.18 to 0.94] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Positive Predictive Value of At-home, CGM-measured Glucose Challenge
Description: Positive predictive value of CGM-glucose 2 hours after at-home glucose beverage ingestion to predict OGTT-2h≥140 mg/dL
Time Frame: 2 Hour Point of Home-OGTT
Measure: Number; unit: percent accuracy of positive tests
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 29
percent accuracy of positive tests | 18.2
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 0.56, 95% CI 2-sided [0.18 to 0.94] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Negative Predictive Value of At-home, CGM-measured Glucose Challenge
Description: Negative predictive value of CGM-glucose 2 hours after at-home glucose beverage ingestion to predict OGTT-2h≥140 mg/dL
Time Frame: 2 Hour Point of Home-OGTT
Measure: Number; unit: percent accuracy of negative tests
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 29
percent accuracy of negative tests | 85.7
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 0.56, 95% CI 2-sided [0.18 to 0.94] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Sensitivity of At-home CGM-measured Fasting Glucose
Description: Sensitivity of baseline CGM-glucose at the time of at-home glucose beverage ingestion to predict fasting OGTT ≥100 mg/dL
Time Frame: 5 Minute Point of Home-OGTT
Population: Of the 35 participants completing the 2-hr CGM-OGTT, 31 had valid data for baseline fasting glucose.
Measure: Number; unit: percentage of true positives
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 31
percentage of true positives | 100
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 1.00 — Area under the receiver operating characteristic curve (AUC) was 1.00 (based on 100% sensitivity) for elevated fasting glucose

8. Secondary Outcome: Specificity of At-home CGM-measured Fasting Glucose
Description: Specificity of baseline CGM-glucose at the time of at-home glucose beverage ingestion to predict fasting OGTT ≥100 mg/dL
Time Frame: 5 Minute Point of Home-OGTT
Population: Of the 35 participants completing the 2-hr CGM-OGTT, 31 had valid data for baseline fasting glucose.
Measure: Number; unit: percentage of true negatives
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 31
percentage of true negatives | 10
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 1.00 — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Positive Predictive Value of At-home CGM-measured Fasting Glucose
Description: Positive predictive value of baseline CGM-glucose at the time of at-home glucose beverage ingestion to predict fasting OGTT ≥100 mg/dL
Time Frame: 5 Minute Point of Home-OGTT
Population: Of the 35 participants completing the 2-hr CGM-OGTT, 31 had valid data for baseline fasting glucose.
Measure: Number; unit: percent accuracy of positive tests
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 31
percent accuracy of positive tests | 3.6
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 1.00 — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Negative Predictive Value of At-home CGM-measured Fasting Glucose
Description: Negative predictive value of baseline CGM-glucose at the time of at-home glucose beverage ingestion to predict fasting OGTT ≥100 mg/dL
Time Frame: 5 Minute Point of Home-OGTT
Population: Of the 35 participants completing the 2-hr CGM-OGTT, 31 had valid data for baseline fasting glucose.
Measure: Number; unit: percent accuracy of negative tests
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 31
percent accuracy of negative tests | 100
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Test type: Other; AUC = 1.00 — [estimate comment as in outcome 7, analysis 1]

11. Other Pre Specified Outcome: Laboratory-measured HbA1c
Description: HbA1c will be measured in the laboratory at baseline to investigate associations with CGM indices obtained during at-home glucose challenge.
Time Frame: Measured at Research Visit
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 39
percent | 5.7 [5.4 to 5.9]
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT fasting glucose and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.3, Spearman correlation; Spearman correlation rho = 0.18
Statistical Analysis 2: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT 2-hour glucose and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.005, Spearman correlation; Spearman correlation rho = 0.50
Statistical Analysis 3: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between delta (difference between fasting and postprandial) home-OGTT glucose and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.01, Spearman correlation; Spearman correlation rho = 0.46
Statistical Analysis 4: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT peak glucose and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.2, Spearman correlation; Spearman correlation rho = 0.23
Statistical Analysis 5: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between time of home-OGTT peak glucose and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.5, Spearman correlation; Spearman correlation rho = 0.14
Statistical Analysis 6: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM mean glucose (mg/dL) and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.1, Spearman correlation; Spearman correlation rho = 0.29
Statistical Analysis 7: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM correlation of variability (CV) and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.4, Spearman correlation; Spearman correlation rho = -0.15
Statistical Analysis 8: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM standard deviation and HbA1c; Test type: Other — Spearman correlation analysis; p = 0.7, Spearman correlation; Spearman correlation rho = -0.06

12. Other Pre Specified Outcome: Laboratory-measured Fasting Glucose
Description: Fasting glucose will be measured in the laboratory at baseline to investigate associations with CGM indices obtained during at-home glucose challenge.
Time Frame: Start of Lab-OGTT
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 39
mg/dL | 84 [80 to 91]
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT fasting glucose and laboratory-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.2, Spearman correlation; Spearman correlation rho = 0.25
Statistical Analysis 2: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT 2-hour glucose and lab-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.3, Spearman correlation; Spearman correlation rho = 0.19
Statistical Analysis 3: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between delta (difference between fasting and postprandial) home-OGTT and lab-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.6, Spearman correlation; Spearman correlation rho = -0.10
Statistical Analysis 4: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT peak glucose and lab-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.3, Spearman correlation; Spearman correlation rho = 0.19
Statistical Analysis 5: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between time of home-OGTT peak glucose and lab-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.6, Spearman correlation; Spearman correlation rho = 0.09
Statistical Analysis 6: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM mean glucose and lab-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.05, Spearman correlation; Spearman correlation rho = 0.35
Statistical Analysis 7: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM coefficient of variability (CV) and lab-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.3, Spearman correlation; Spearman correlation rho = -0.18
Statistical Analysis 8: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM standard deviation (SD) and lab-OGTT fasting glucose; Test type: Other — Spearman correlation analysis; p = 0.7, Spearman correlation; Spearman correlation rho = -0.07

13. Other Pre Specified Outcome: Laboratory-measured 2-hour Glucose
Description: 2-hour OGTT glucose will be measured in the laboratory at baseline to investigate associations with CGM indices obtained during at-home glucose challenge.
Time Frame: 2 Hour Point of Lab-OGTT
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | CGM Use for T2D Risk Evaluation
Number analyzed (Participants) | 39
mg/dL | 112 [101 to 126]
Statistical Analysis 1: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT fasting glucose and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.6, Spearman correlation; Spearman correlation rho = 0.10
Statistical Analysis 2: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT 2-hour glucose and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.1, Spearman correlation; Spearman correlation rho = 0.31
Statistical Analysis 3: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between delta (difference between fasting and postprandial) home-OGTT glucose and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.2, Spearman correlation; Spearman correlation rho = 0.25
Statistical Analysis 4: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between home-OGTT peak glucose and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.2, Spearman correlation; Spearman correlation rho = 0.26
Statistical Analysis 5: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between time of home-OGTT peak glucose and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.2, Spearman correlation; Spearman correlation rho = 0.27
Statistical Analysis 6: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM mean glucose and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.08, Spearman correlation; Spearman correlation rho = 0.31
Statistical Analysis 7: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM coefficient of variability (CV) and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.4, Spearman correlation; Spearman correlation rho = 0.15
Statistical Analysis 8: Comparison: CGM Use for T2D Risk Evaluation; Correlation analyses were performed to assess the relationship between CGM standard deviation (SD) and lab-OGTT 2-hour glucose; Test type: Other — Spearman correlation analysis; p = 0.1, Spearman correlation; Spearman correlation rho = 0.28

ADVERSE EVENTS:
Time Frame: Adverse event information was collected for the study duration of 10 days.
Arm/Group | CGM Use for T2D Risk Evaluation
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 3/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CGM Use for T2D Risk Evaluation (N=39)
Rash due to CGM adhesive (Skin and subcutaneous tissue disorders) | 2
Emesis due to OGTT beverage (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT05404711/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT05404711/ICF_000.pdf